CLINICAL TRIAL: NCT05727553
Title: Implementation of Online Adaptive Radiotherapy for Breast Cancer Patients on Ethos
Brief Title: Implementation of Online Adaptive Radiotherapy for Breast Cancer Patients on Ethos (BREAST-ART)
Acronym: BREAST-ART
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, H.J.G.D. van den Bongard, Principal Investigator, Amsterdam UMC, location VUmc
Other Study IDs: IRB00002991
Record Dates: First submitted 2022-12-13; First posted 2023-02-14 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Radiotherapy; Online adaptive; Postoperative
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast cancer patients: Breast cancer patients treated with postoperative radiotherapy in an online adaptive workflow on Ethos.
  Interventions: Radiation: Online adaptive radiotherapy

INTERVENTIONS:
Radiation: Online adaptive radiotherapy — Postoperative radiotherapy will be indicated conform the standard medical care and guidelines. The radiation is delivered with online adaptive radiotherapy performed on the Ethos. This technique will be evaluated.

SUMMARY:
Postoperative radiotherapy is for the majority of breast cancer patients the standard of care. During postoperative radiotherapy, unexpected dosimetric deviations can occur due to breast contour changes resulting from resorption of postoperative breast or chest wall seroma/hematoma, oedema either postoperatively or during irradiation, or arm/body positioning variation. In approximately 10% of cases, repositioning after setup imaging is not sufficient, and offline plan adaptation is required. When a new treatment planning is required in the standard offline workflow this will take in general 2 days. By using an online adaptive workflow with a daily treatment planning this delay and extra work caused by offline plan adaptation can be omitted. The aim of this study is to translate the offline adaptive workflow to an online adaptive workflow, and investigate the experiences of patients who have been treated with online adaptive radiotherapy for breast cancer (BREAST-ART).

DETAILED DESCRIPTION:
In this single-arm prospective BREAST-ART study breast cancer patients with an indication for postoperative radiotherapy will be treated according to the Dutch and institutional guidelines. Target volumes will be the whole breast, chest wall, axillary levels, tumor bed boost and partial breast irradiation on the right side and left side with a deep inspiration breath hold technique. Robust templates are developed for offline and online treatment planning with an IMRT tangential multiple-beam setup. A simulation of the online adaptive workflow is performed in breast cancer patients already treated on the Ethos-linac with the standard offline adaptive workflow. Patients will be treated following the online adaptive workflow delivered on the Ethos-Linac. Patient experience will be evaluated using an in-house developed questionnaires after the first and last fraction, scoring treatment satisfaction on a 4-point Likert scale. Furthermore, all dosimetric data, volume details, DICOM images and the time spend on all parts of the online adaptive workflow will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients referred for postoperative radiotherapy of the breast, chest wall, axillary levels, tumor bed boost or partial breast irradiation.
* Age of 18 years and older.
* Adequate understanding and communicating the Dutch language.
* Written informed consent for use of routinely collected clinical data and to fill out questionnaires.

Exclusion Criteria:

* Patients not suitable for postoperative radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients undergoing postoperative radiation treatment.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Time spend on the online adaptive workflow | 30 minutes
  All separate parts of the online adaptive workflow will be registered in minutes, starting when the patients enters the room of the radiation machine until the patient leaves the room.
Patient experience | 10 minutes
  Patient experience is measured using an in-house designed short study questionnaire after the first and the last radiation fraction. The questionnaires is on a 4-point Likert scale with a lowest score for discomfort and the highest score appears for good comfort.
Dosimetric data | 1 week
  The dosimetric data of the standard offline treatment plan (reference plan), scheduled plan and the online adapted treatment plan (adapted plan) will be compared.
DICOM images | 1 week
  DICOM images of the standard offline treatment plan (reference plan), scheduled plan and the online adapted treatment plan (adapted plan) will be compared.
Volumes | 1 week
  Target volumes of clinical target volume (CTV), planning target volume (PTV), coverage of CTV and PTV will be registred in cubic centimetres.
Number of monitor units (MU). | 1 week
  The number of monitor units (MU) will be compared between the reference treatment plan, scheduled plan and adapted treatment plan.

SECONDARY OUTCOMES:
Radiation associated toxicity | Baseline, 1 month and 3 months after radiotherapy
  Toxicity will be assessed by the Common Terminology Criteria Adverse Events version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Desirée van den Bongard, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No